CLINICAL TRIAL: NCT07323342
Title: Evaluation of the Efficacy and Safety of Intra-Articular Hyaluronic Acid Combined With Fibrinogen in Patients With Knee Osteoarthritis
Brief Title: Effectiveness and Safety of Intra-Articular Hyaluronic Acid Combined With Fibrinogen in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cao Kim Xoa (Other)
Responsible Party: Sponsor-Investigator, Cao Kim Xoa, PhD Candidate, Clinical Pharmacology, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24295 - ĐHYD; 24295-DHYD (Other: University of Medicine and Pharmacy at Ho Chi Minh City (UMP))
Record Dates: First submitted 2025-12-16; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Hyaluronic acid; Intra-articular injection; Pain management
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a single-arm interventional study in which all participants receive intra-articular hyaluronic acid combined with fibrinogen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-articular combination Hyaluronic Acid and Fibrinogen (Experimental): Participants with knee osteoarthritis receive intra-articular injections of hyaluronic acid combined with fibrinogen according to routine clinical practice. This is a single-arm, post-marketing study evaluating effectiveness and safety outcomes.
  Interventions: Device: Intra-articular hyaluronic acid combined with fibrinogen

INTERVENTIONS:
Device: Intra-articular hyaluronic acid combined with fibrinogen — Participants with knee osteoarthritis receive intra-articular injections of hyaluronic acid combined with fibrinogen as part of routine clinical practice. The intervention is administered according to standard post-marketing use. This single-arm study evaluates the effectiveness and safety of the intervention without a comparator.

SUMMARY:
This study aims to evaluate the effectiveness and safety of intra-articular injections of hyaluronic acid combined with fibrinogen in patients with knee osteoarthritis.

Knee osteoarthritis is a common degenerative joint disease that causes pain, stiffness, and reduced mobility, significantly affecting quality of life. Hyaluronic acid injections are widely used to relieve symptoms, but their effectiveness may be limited in some patients. Fibrinogen has potential biological effects that may enhance tissue repair and anti-inflammatory responses.

In this single-arm clinical study, patients with knee osteoarthritis will receive intra-articular injections of a combination of hyaluronic acid and fibrinogen. Clinical outcomes, including pain relief, functional improvement, and adverse events, will be assessed during follow-up visits.

The results of this study may provide additional evidence regarding the potential benefits and safety of combining hyaluronic acid with fibrinogen for the treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
This is a prospective, single-arm clinical study designed to evaluate the efficacy and safety of intra-articular hyaluronic acid combined with fibrinogen in patients with knee osteoarthritis.

Eligible patients diagnosed with knee osteoarthritis according to clinical and radiographic criteria will be enrolled. All participants will receive intra-articular injections of a combination of hyaluronic acid and fibrinogen administered under sterile conditions.

The primary objectives of the study are to assess changes in pain intensity and knee function following treatment. Secondary objectives include evaluation of functional outcomes, patient-reported quality of life, and the occurrence of adverse events related to the intervention.

Patients will be followed for a predefined period after injection, during which clinical assessments will be performed at scheduled visits. Pain and functional outcomes will be evaluated using validated clinical scales. Safety assessments will include monitoring and recording of any local or systemic adverse events throughout the study period.

This study is conducted as part of a doctoral research project in clinical pharmacology at the University of Medicine and Pharmacy at Ho Chi Minh City. The study protocol has been reviewed and approved by the Institutional Review Board of the University of Medicine and Pharmacy at Ho Chi Minh City prior to initiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 45 to 75 years.
* Diagnosed with primary knee osteoarthritis according to the American College of Rheumatology (ACR) 1991 criteria.
* Vietnamese patients.
* Patients who have provided written informed consent to participate in the study.
* Patients with full-length standing lower limb radiographs showing a mechanical axis deviation of less than 10 degrees.
* Body mass index (BMI) between 18.5 and 35 kg/m².

Exclusion Criteria:

* Active joint infection or systemic infection.
* Presence of other joint diseases such as rheumatoid arthritis, gout, malignancy-related joint disease, or significant knee trauma.
* Acute concomitant medical conditions such as high fever, acute myocardial infarction, or pneumonia.
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) within 10 days prior to enrollment or intra-articular corticosteroid injection within 3 months before enrollment.
* Presence of knee joint effusion at the time of screening.
* History of hypersensitivity or allergy to hyaluronic acid.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in WOMAC total score | Baseline, 2 weeks, 1 month, 3 months, 6 months, and 12 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score is used to assess pain, stiffness, and physical function in patients with knee osteoarthritis. Scores range from 0 to 96, with higher scores indicating worse symptoms.
Change from baseline in pain intensity at rest measured by Visual Analog Scale (VAS) | Baseline, 2 weeks, 1 month, 3 months, 6 months, and 12 months
  Pain intensity at rest is assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.
Change from baseline in pain intensity during movement measured by Visual Analog Scale (VAS) | Baseline, 2 weeks, 1 month, 3 months, 6 months, and 12 months
  Pain intensity during movement is assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.

SECONDARY OUTCOMES:
Change from baseline in Lysholm Knee Scoring Scale | Baseline, 3 months, 6 months, and 12 months
  The Lysholm Knee Scoring Scale is used to assess knee function. Scores range from 0 to 100, with higher scores indicating better knee function.
Change from baseline in physical health measured by SF-36 Physical Component Summary (PCS) | Baseline, 3 months, 6 months, and 12 months
  Physical health-related quality of life is assessed using the Short Form-36 Health Survey (SF-36) Physical Component Summary (PCS). Scores range from 0 to 100, with higher scores indicating better physical health.
Change from baseline in mental health measured by SF-36 Mental Component Summary (MCS) | Baseline, 3 months, 6 months, and 12 months
  Mental health-related quality of life is assessed using the Short Form-36 Health Survey (SF-36) Mental Component Summary (MCS). Scores range from 0 to 100, with higher scores indicating better mental health.
Radiographic severity of knee osteoarthritis assessed by Kellgren-Lawrence grading system | Baseline and 12 months
  Radiographic severity of knee osteoarthritis is assessed using standard knee X-ray and graded according to the Kellgren-Lawrence grading system (Grade 0-4), with higher grades indicating more severe osteoarthritis.
Incidence of adverse events following intra-articular hyaluronic acid-fibrinogen injection | From baseline up to 12 months after intra-articular injection
  Safety is assessed by the incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) related to intra-articular injection of hyaluronic acid combined with fibrinogen. Adverse events include local reactions such as pain, swelling, joint effusion, and infection, as well as systemic adverse events occurring during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Anh Tang Ha, MD, PhD, Principal Investigator — Xuong Khop Viet Clinic; Manh Hung Tran, PhD, Principal Investigator — Head, Department of Pharmacology, School of Pharmacy, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam
Locations (1):
- Xuong Khop Viet clinic, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Han SB, Seo IW, Shin YS. Intra-Articular Injections of Hyaluronic Acid or Steroids Associated With Better Outcomes Than Platelet-Rich Plasma, Adipose Mesenchymal Stromal Cells, or Placebo in Knee Osteoarthritis: A Network Meta-analysis. Arthroscopy. 2021 Jan;37(1):292-306. doi: 10.1016/j.arthro.2020.03.041. Epub 2020 Apr 17. PMID 32305424
- [Result] David BM, Madsen BW, Ilett KF. Plasma binding of disopyramide. Br J Clin Pharmacol. 1980 Jun;9(6):614-8. doi: 10.1111/j.1365-2125.1980.tb01090.x. No abstract available. PMID 7387819